CLINICAL TRIAL: NCT04808128
Title: The Effect of Energy Drinks Consumption on Acute Physiological and Psychological Responses of Israeli Arab Adolescents: In Search for a Possible Microbiota-derived Metabolite-dependent Mechanism.
Brief Title: The Effect of Energy Drinks Consumption on Acute Physiological and Psychological Responses of Israeli Arab Adolescents
Acronym: EDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Hai College (Other)
Collaborators: Saint Vincent De Paul - French Hospital - Nazareth (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TelHaiC-EDE
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Energy Drinks
Keywords: Energy drinks (EDs); Blood pressure (BP); Glucose tolerance; Metabolite profiles; Mood; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Drink A + SC (Experimental): In t0 the group will receive 250 ml XL energy drink + 20 gr sucrose.
  Interventions: Other: Drink A + SC
- Drink B + SC (Active Comparator): In t0 the group will receive 250 ml Fanta soft drink + 20 gr sucrose.
  Interventions: Other: Drink B + SC
- Drink C + SC (Active Comparator): In t0 the group will receive 250 ml soda water + 47 gr sucrose.
  Interventions: Other: Drink C + SC
- Drink A + CC (Experimental): In t0 the group will receive 250 ml XL energy drink + 20gr complex carbohydrates from one slice of bread (30g) and one spoon of hummus.
  Interventions: Other: Drink A + CC
- Drink B + CC (Active Comparator): In t0 the group will receive 250 ml Fanta soft drink + 20gr complex carbohydrates from one slice of bread (30g) and one spoon of hummus.
  Interventions: Other: Drink B + CC
- Drink C + CC (Active Comparator): In t0 the group will receive 250 ml soda water + 27gr sucrose + 20gr complex carbohydrates from one slice of bread (30g) and one spoon of hummus.
  Interventions: Other: Drink C + CC

INTERVENTIONS:
Other: Drink A + SC — Consumption of energy drink that contains 80mg caffeine and 27g carbohydrates per 250ml together with simple carbohydrates.
  Arms: Drink A + SC
Other: Drink B + SC — Consumption of soft drink, non-caffeine drink that contains 27g carbohydrates per 250ml together with simple carbohydrates.
  Arms: Drink B + SC
Other: Drink C + SC — Consumption of soda water, non-caffeine and non-carbohydrate drink together with simple carbohydrates.
  Arms: Drink C + SC
Other: Drink A + CC — Consumption of energy drink that contains 80mg caffeine and 27g carbohydrates per 250ml together with complex carbohydrates.
  Arms: Drink A + CC
Other: Drink B + CC — Consumption of soft drink, non-caffeine drink that contains 27g carbohydrates per 250ml together with complex carbohydrates.
  Arms: Drink B + CC
Other: Drink C + CC — Consumption of soda water, non-caffeine and non-carbohydrate drink together with complex carbohydrates.
  Arms: Drink C + CC

SUMMARY:
Quasi-experiment and Cross-sectional study, six-arm design protocol will be carried out. The study will be conducted under the Declaration of Helsinki.

The current study will assess the effects of EDs consumption on the physiological and psychological responses of Israeli Arab adolescents. These effects will also be examined in association with the adolescent's plasma metabolite profiles.

The study has five specific aims: (1) to assess the effects of ED consumption with or without a meal, on Israeli Arab adolescents glucose levels by using mixed meal tolerance test (MMTT) (2) to assess the effect of ED consumption with or without a meal on their blood pressure (3) to evaluate the association between ED consumption per day by the Israeli Arab adolescents and their nutritional status and habits (4) to examine for possible associations between Israeli Arab adolescents psychological status (i.e. mood and anxiety) and ED consumption per day (5) to examine for possible associations between ED and caffeine consumption and plasma metabolite profiles and, the subject's psychological status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Israeli Arab adolescents
* aged 14.5-17.5 years

Exclusion Criteria:

* diabetes
* hypoglycemic episodes
* coronary heart disease, cardiac arrhythmia, secondary hypertension, structural heart lesions
* hepatic or renal disorders
* autonomic neuropathy
* epilepsy
* obstructive sleep apnea
* migraines
* caffeine intolerance
* eating disorders or other mental disorders or those with prescribed psychiatric medications

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Blood sugar change | First measurement at baseline, before consuming the meal, and four times during the intervention - 15, 30, 60 and 120 minutes after consuming the meal
  Change in blood sugar levels (mg/dL) will be measured with the mixed meal tolerance test (MMTT) five times - one time at baseline (before consuming the meal) and four times during the intervention (15, 30, 60 and 120 minutes after consuming the meal).
Anxiety status | During the intervention, 60 minutes after consuming the meal.
  Anxiety status will be measured one time during the intervention - 60 minutes after consuming the meal, with the SCARED-R questionnaire (Muris et al., 1999) in Arabic. SCARED-R is a self-report questionnaire which measures anxiety status in the last 3 months. Contains 41 statements (such as "I am nervous") in Likert scale of 0 ("Not True or Hardly Ever True") to 2 ("Very True or Often True"). A total score of ≥ 25 may indicate the presence of an Anxiety Disorder.
Mood change | First measurement at baseline, before consuming the meal, and another measurement during the intervention, 60 minutes after consuming the meal.
  Mood change will be measured two times - one time at baseline (before consuming the meal) and another time during the intervention - 60 minutes after consuming the meal. Mood will be measured with the UMACL questionnaire (Matthews et al., 1990) in Arabic. UMACL is a self-report questionnaire which measures the current mood of the subject. Contains 29 statements (such as "I am happy"), in Likert scale of 1 ("absolutely") to 4 ("not at all"). The higher the score, the better the current mood is.
Insulin levels status | During the intervention, between 30-45 minutes after consuming the meal.
  Insulin levels status will be measured based on blood samples that will be taken from subjects during the intervention, 30-45 minutes after consuming the meal. Analysis will take place after the data collection stage.
SCFA levels status | During the intervention, between 30-45 minutes after consuming the meal.
  SCFA levels status will be measured based on blood samples that will be taken from subjects during the intervention, 30-45 minutes after consuming the meal. Analysis will take place after the data collection stage.
HR change | First measurement at baseline, before consuming the meal, and four times during the intervention - 15, 30, 60 and 120 minutes after consuming the meal
  Changes in heart rate (BPM) will be measured five times - First at baseline (before consuming the meal) and four times during the intervention - 15, 30, 60 and 120 minutes after consuming the meal.

SECONDARY OUTCOMES:
BP change | First measurement at baseline, before consuming the meal, and four times during the intervention - 15, 30, 60 and 120 minutes after consuming the meal
  Changes in systolic and diastolic blood pressure (mm Hg) will be measured five times - one time at baseline (before consuming the meal) and four times during the intervention (15, 30, 60 and 120 minutes after consuming the meal).
Life habits status | During intervention, 60 minutes after consuming the meal.
  Life habits status will be measured one time during the intervention, 60 minutes after consuming the meal, using the Nutritional Status Questionnaire (based on the Israeli Ministry of Health 2nd nutrition survey [MABAT], 2017) in Arabic. The questionnaire includes 8 questions (such as "Are you eating breakfast?"), with no cut-off score.
Energy drinks consumption status | During intervention, 60 minutes after consuming the meal.
  Energy drinks consumption status will be measured one time during the intervention, 60 minutes after consuming the meal, using a questionnaire by Attila & Çakir, 2011, in Arabic. The questionnaire includes 9 questions (such as "Do you drink energy drinks?"), with no cut-off score.
Caffeine consumption frequency | During intervention, 60 minutes after consuming the meal.
  Caffeine consumption frequency will be measured one time during the intervention, 60 minutes after consuming the meal, using a questionnaire from Harpaz et al., 2016 in Arabic. The questionnaire contains 2 questions (such as "Please choose the products you consumed during the last week"), with no cut-off score.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Nimri, Dr., Principal Investigator — Nutritional sciences Department Tel-Hai College
Locations (1):
- Saint Vincent De Paul hospital, Nazareth, Israel

IPD SHARING:
Plan to Share IPD: No